CLINICAL TRIAL: NCT01567319
Title: Biological Standardization of D. Glomerata, L. Perenne, S. Cereale and O. Europaea Pollen Extracts in Patients Sensitized to Them.
Brief Title: Biological Standardization of D. Glomerata, L. Perenne, S. Cereale and O. Europaea Pollen Extracts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BIA-STD-002; 2011-001270-25 (EudraCT Number)
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Sensitization to Allergens
Keywords: Sensitization; Skin Prick Test; Standardization; sources of: D. glomerata, L. perenne, S. cereale and O. europaea
MeSH Terms: interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Allergic Subjects (Experimental)
  Interventions: Biological: Skin Prick Test
- Atopic Subjects (Active Comparator): Patients sensitized to other allergenic sources but the allergen extracts under investigation.
  Interventions: Biological: Skin Prick Test - Atopic Subjects
- No Atopic Subjects (Active Comparator): Healthy volunteers.
  Interventions: Biological: Skin Prick Test - No Atopic Subjects

INTERVENTIONS:
Biological: Skin Prick Test — Skin prick test of 4 concentrations of each allergenic source, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm. Assessment of the wheal size after 15 minutes.
  Arms: Allergic Subjects
Biological: Skin Prick Test - Atopic Subjects — Skin prick test of 4 concentrations of each allergenic source,together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm. Assessment of the wheal size after 15 minutes.
  Arms: Atopic Subjects
Biological: Skin Prick Test - No Atopic Subjects — Skin prick test of 4 concentrations of each allergenic source, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every subjects in duplicate on the volar surface of the forearm. Assessment of the wheal size after 15 minutes.
  Arms: No Atopic Subjects

SUMMARY:
Allergen extracts are complex mixtures of proteins and contain varying amounts of allergenic and non-allergenic components. Many factors such as the biovariability, differences in extraction process and subsequent handling of allergens can affect the final composition, potency, and stability of allergen preparations. Genetic diversity of affected people adds another level of complexity. In order to control variability and to achieve consistency and reproducibility for optimal safety and sensitivity/specificity, it is essential to standardize the amount of allergen used in prick tests. Therefore, the system for biological standardization mainly used in Europe still is the biological calibration of in-House Reference Preparations (IHRP). The method has been adopted by the Nordic Council on Medicines as the Nordic Biological Unit, Histamine Equivalent Potency (HEP) or Skin Prick Test (SPT) value. The aim of this procedure is to estimate the biological activity of allergen extracts. The activity of an allergen extract is defined as 1 SPT per ml, when the extract provokes a specific skin reaction with a wheal of the same size as a wheal provoked by reference histamine at a concentration of 10 mg/ml, when both solutions are administrated using the same technique (prick testing) on at least 20 individuals who are sensitized to the allergen concerned.

The present study aims to standardize the allergen extracts of Dactylis glomerata, Lolium perenne, Secale cereale y Olea europaea by using this method.

ELIGIBILITY:
Inclusion Criteria:

A. Subjects sensitized to one or more allergen extracts:

1. Positive clinical history with inhalant allergy to at least one of the allergen to be standardized.
2. At least one positive prick test (mean wheal diameter greater or equal than 3mm) .
3. Positive prick test (wheal diameter greater or equal to 3 mm) to Histamine 10 mg/ml
4. Age: 18-60 years
5. Written informed consent
6. Patients will preferably be monosensitized, or with clinically relevant sensitization , or with primary sensitization (maximum cutaneous reactivity) to the extracts under investigation.
7. Women of child-bearing potential must have a negative urine pregnancy test at the time they begin the study.

B. Atopic Subjects:

1. Age: 18-60 years
2. Written informed consent
3. Positive prick test (wheal diameter greater or equal to 3 mm) to Histamine 10 mg/ml
4. Negative prick test (mean wheal diameter less or equal to 3mm) when tested with already standardized extracts of the allergens under investigation or with cross reactive extracts.
5. Women of child-bearing potential must have a negative urine pregnancy test at the time they begin the study.

C. No Atopic Subjects:

1. Age: 18-60 years.
2. Written informed consent
3. Positive prick test (wheal diameter greater or equal to 3 mm) to Histamine 10 mg/ml
4. Negative prick test (mean wheal diameter less or equal to 3mm)to all allergens tested in diagnostic prick test.
5. Women of child-bearing potential must have a negative urine pregnancy test at the time they begin the study.

Exclusion Criteria (shared by the 3 groups):

1. Immunotherapy in the 2 years prior to the study against either the allergen to be tested or an allergen which is cross-reactive. (it is not applicable to no atopic patients)
2. Any drug which may interfere with the cutaneous test or with its result.
3. Any medical condition that from investigator's point of view the skin prick test cannot be done .
4. Women who are pregnant or breast-feeding or are child-bearing age and who have not demonstrated that they have been surgically sterilized or have other means of not bearing children.

4.Subjects who have participated in another clinical trial within 3 months prior to this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Wheal size area | 15 minutes after skin prick test
  The primary efficacy variable will be the wheal size area at the site of the puncture of the immediate phase reaction in mm2.

CONTACTS AND LOCATIONS:
Overall Officials: Arantza Vega, MD, Principal Investigator — Hospital Universitario de Guadalajara; Pilar Alba, MD, Principal Investigator — Hospital de Manises; José Manuel Zubeldia, MD, Principal Investigator — Hospital Universitario Gregorio Marañón; María Ángeles Gonzalo Garijo, MD, Principal Investigator — Hospital Universitario Infanta Cristina; Carlos Colás, MD, Principal Investigator — Hospital Clínico Universitario Lozano Blesa; Blanca Saenz de San Pedro, Principal Investigator — Complejo Hospitalario de Jaén; Lourdes Fernández, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (7):
- Spain (7):
  - Hospital de Manises, Manises, Valencia
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza